CLINICAL TRIAL: NCT06351956
Title: New Onset Cardiac Arrhythmias in Septic Patients in Critical Care Setting, Predictors and Outcomes.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Sameh Anwer, Resident, Assiut University
Other Study IDs: Arrhythmias in Septic Patients
Record Dates: First submitted 2024-03-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrhythmia
Keywords: cardiac arrhythmia; sepsis; critical care
MeSH Terms: conditions — Arrhythmias, Cardiac; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New Onset Cardiac Arrhythmias in Septic Patients in Critical Care Setting, Predictors and Outcomes

DETAILED DESCRIPTION:
Sepsis is recently defined as life-threatening condition caused by dysregulated body response to infection leading to organ dysfunction and even death. Patients who are vulnerable to catch sepsis are those with immune-compromising diseases, old aged people and chronic medical condition such as diabetes, chronic kidney diseases or cancer. Sepsis is symptomized by fever or hypothermia, tachycardia, tachypnea. In critical care units, septic patient are predisposed to have different cardiovascular manifestation as atrial fibrillation, atrial flutter, hypotension, etc. . Many studies reported the association between atrial fibrillation and septic patients in critical care as a complication of sepsis; but data regarding factors and fates is still insufficient. So in this study we aim to observe critical ill patients with sepsis to assess and evaluate the predisposing factors leading to new onset of cardiac arrhythmia in septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient of 18 years old and above of both gender admitted with manifestation of sepsis.

Exclusion Criteria:

* Patients below 18 years old.
* Pregnant females.
* Patients with cardiac arrhythmia before admission in the critical unit.
* Patients with previous cardiac surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged from 18 years and above of both sexes (male and female) who are admitted in critical care unit in Assuit University Hospital and diagnosed by sepsis will be enrolled if matched the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk Factors of cardiac arrhythmias in septic patients in CU. | 3 week from admission in CU
  any medical condition precipitate the occurrence of cardiac arrhythmia
Fates of cardiac arrhythmia. | 1 month from the primary endpoint
  what complications will precipitate the arrhythmia or the recovery achievement

SECONDARY OUTCOMES:
The frequent type of arrhythmias. | 2 years from starting collaboration
  the most frequent type of cardiac arrhythmia
Mortality rate due to new onset arrhythmia. | 2 years from starting collaboration
  the number of deaths from the enrolled patients

REFERENCES:
- [Result] Marik PE, Taeb AM. SIRS, qSOFA and new sepsis definition. J Thorac Dis. 2017 Apr;9(4):943-945. doi: 10.21037/jtd.2017.03.125. No abstract available. PMID 28523143
- [Result] Makrygiannis SS, Margariti A, Rizikou D, Lampakis M, Vangelis S, Ampartzidou OS, Katsifa K, Tselioti P, Foussas SG, Prekates AA. Incidence and predictors of new-onset atrial fibrillation in noncardiac intensive care unit patients. J Crit Care. 2014 Aug;29(4):697.e1-5. doi: 10.1016/j.jcrc.2014.03.029. Epub 2014 Apr 4. PMID 24814972